CLINICAL TRIAL: NCT06993129
Title: A Multi-Site Hybrid Type I Effectiveness-Implementation Randomized Trial of an Emergency Care Action Plan for Infants With Medical Complexity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Christian Pulcini, Assistant Professor of Emergency Medicine and Pediatrics, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FP00005878
Record Dates: First submitted 2025-05-12; First posted 2025-05-28 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Chronic Disease Management; Infants Health; Emergency; Utilization, Health Care; Caregiver Stress
Keywords: Children with Medical Complexity; Hybrid Implementation Trial; Health Service Utilization
MeSH Terms: conditions — Emergencies; Patient Acceptance of Health Care; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emergency Care Action Plan (Experimental): An Emergency Care Action Plan (ECAP) is a brief, pre-populated summary of suggested emergency management for children with medical complexity, embedded in the electronic health record.
  Interventions: Other: Emergency Care Action Plan
- Standard Care (No Intervention): The current standard of care does not include emergency care planning.

INTERVENTIONS:
Other: Emergency Care Action Plan — An Emergency Care Action Plan (ECAP) is a brief, pre-populated summary of suggested emergency management for children with medical complexity, embedded in a patient's electronic health record for access by providers in an emergency. Patients/families will have digital access to the ECAP and be given a paper copy. The patient's care team and caregiver(s) (parent/legal guardian) will collaborate to create an individualized ECAP containing the following content: caregiver contact information, patient summary, anticipated emergency presentations with suggested management, problem list (emergency relevant only), medication list, technology dependence, baseline important physical exam findings, baseline vital signs, allergies, advance directive information, contact information for established care providers, and other important information.
  Arms: Emergency Care Action Plan

SUMMARY:
Infants with medical complexity (IMC) are a challenging population with more emergency department visits, inpatient stays, and higher healthcare costs than other children. IMC also experience lower quality emergency health care. The PI and team propose to adapt and put into place an emergency care action plan (ECAP) for IMC across four US hospitals, working directly with medical providers and families in each setting. After the tool is made available to providers and families, the PI and team will measure if the ECAP tool helps decrease the number of hospitalizations (primary research outcome) for IMC, as well as if the ECAP is feasible, acceptable, and useable for those using the ECAP over a one-year period.

DETAILED DESCRIPTION:
The project goal is to optimize and implement an emergency care action plan (ECAP) developed previously by the PI and team (through an NIH K23 award) to improve emergency care for infants with medical complexity, a particularly challenging subset of CMC with high utilization and unique challenges in the acute care setting. Dr. Pulcini and team will conduct a hybrid type I effectiveness-implementation randomized trial of the ECAP at four sites (Children's Hospital Colorado, Cincinnati Children's Hospital Medical Center, Children's Hospital of Philadelphia, and the University of Vermont), measuring both health care outcomes/effectiveness (primary endpoint: number of hospitalizations) and implementation (endpoints include acceptability, feasibility, and useability). Dr. Pulcini and team will also measure key secondary health service measures (ex. ED visits, caregiver stress and self-efficacy) and monitor facilitators and barriers to implementation throughout the trial at each site.

ELIGIBILITY:
Inclusion Criteria:

* Age 0 to 6 months
* Admitted to the University of Vermont Medical Center, Cincinnati Children's Hospital, Children's Hospital of Philadelphia, or Colorado Children's Hospital Neonatal Intensive Care Unit (NICU),
* Meets or is expected to meet Children with Medical Complexity status as determined by the treating NICU clinician and defined as "children with multiple significant chronic health problems including multiple organ systems, which result in functional limitations, high health care needs or utilization, and often require need for, or use of, medical technology."
* Has three or more documented complex chronic conditions (CCCs)

Exclusion Criteria:

* Does not have a caregiver participant who agrees to their participation in the study to complete follow-up surveys
* Does not intend to use the hospital or affiliated sites of which they were recruited from for care during the one-year trial period

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Hospitalization | Day 0 (NICU discharge) to Month 12
  Dichotomous variable for hospitalization vs. no hospitalization (yes/no)

SECONDARY OUTCOMES:
Number of ED Visits | Day 0 (NICU discharge) to Month 12
  Number of ED visits
Usability | Day 0 (NICU discharge) to Month 12
  Will assess usability using an adaption of the System Usability Scale (SUS) and qualitative assessment of implementation barriers and facilitators (for intervention group only).
Acceptability | Day 0 (NICU discharge) to Month 12
  Will assess acceptability using an adaptation of the Theoretical Framework of Acceptability (TFA), including the following constructs: affective attitude, burden, intervention coherence, self-efficacy, and opportunity costs. Qualitative assessment of implementation barriers and facilitators (for intervention group only) will also elicit perspectives of acceptability.
Feasibility of Intervention | Day 0 (NICU discharge) to Month 12
  Will assess feasibility using an adaptation of the Feasibility of Intervention Measure (FIM), as well as a qualitative assessment of implementation barriers and facilitators (for intervention group only).

OTHER OUTCOMES:
Caregiver Stress | Day 0 (NICU discharge) to Month 12
  Will measure caregiver self-perceived stress and compare between the intervention and standard care by using the University of Washington Caregiver Stress Scale 3-Item Short Form.
Caregiver Self-Efficacy | Day 0 (NICU discharge) to Month 12
  Will measure caregiver self-efficacy and compare between the intervention and standard care by using an adaptation of the Parent Measure of Self-Efficacy Managing a Child's Medications and Treatments, including assessment of self-efficacy in two domains: (1) healthcare information and decision-making, and (2) symptoms identification and management.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Colorado Children's Hospital, Aurora, Colorado
  - Cincinnati Children's Hospital and Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Vermont Medical Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after de-identification will be shared (text, tables, figures and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 26 months following article publication.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research for individual participant data meta analysis. Proposals may be submitted up to 36 months following article publication. Proposals must be reviewed and approved by an independent review committee identified for this purpose. Proposals should be directed to Christian.Pulcini@uvm.edu.

REFERENCES:
- [Background] Pulcini CD, Broder-Fingert S, Callas P, Dayan PS, Drath B, Gravel-Pucillo C, Kuo DZ, Lamberson M, Mistry RD, Palaza A, Stevens M, Yeager J, Stapleton RD. Human-Centered Design to Create an Emergency Care Action Plan for Children With Medical Complexity. Pediatrics. 2025 Feb 12:e2024069125. doi: 10.1542/peds.2024-069125. Online ahead of print. PMID 39933576